CLINICAL TRIAL: NCT01080157
Title: An Evaluation of a Noninvasive Diabetes Screening Device in Subjects at Risk for Diabetes
Brief Title: Evaluation of a Noninvasive Diabetes Screening Device in Subjects at Risk for Diabetes
Acronym: ENGINE
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2712
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes
Keywords: Diabetes; Diabetes Screening; Experimental Medical Device
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteers 18+, at risk for diabetes
  Interventions: Device: SCOUT DS measurement

INTERVENTIONS:
Device: SCOUT DS measurement — Non-invasive 3-5 volar forearm scan

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the SCOUT DS in measuring the concentration of substances (advanced glycation endproducts) in the skin. These substances have been found to be in higher concentrations in people with diabetes and high blood sugar. The SCOUT DS is being developed to help doctors measure these substances in skin and possibly help doctors diagnose diabetes.

DETAILED DESCRIPTION:
The trial will be a prospective, multi-center, paired data, cohort screening trial. Up to 960 subjects will complete the study to determine the relative accuracy of SCOUT DS compared to the FPG and HbA1c tests in screening for abnormal glucose tolerance. All methods will be compared to the 2 hour value of the OGTT. An algorithm utilizes skin optical modeling as well as the spectral and blood assay data accumulated from the initial phase of the study to produce a risk score for abnormal glucose tolerance. This algorithm and the calculation of the score will be integrated into the SCOUT DS for prospective testing. The design requires three patient visits to the clinical site and up to a total of seven measurements on the SCOUT device.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 45 years; OR
2. Age 18 to 44 years and a BMI > 25 kg/m² with one or more of the following risk factors:

   * Elevated waist circumference, > 35 inches for women and >40 inches for men
   * Habitually physically inactive (does not exercise regularly)
   * Has a first-degree relative with diabetes
   * African American, Latino, Native American, Asian American, Pacific Islander
   * Has delivered a baby weighing > 9 lb or diagnosed with gestational diabetes
   * Hypertension (≥130/≥ 85 mmHg) or being treated for hypertension
   * HDL cholesterol level < 35 mg/dL and/or a fasting triglyceride level ≥ 250 mg/dL or being treated for dyslipidemia with medication
   * Has been previously diagnosed with Polycystic Ovary Syndrome (PCOS)
   * Had impaired glucose tolerance or impaired fasting glucose on previous testing within the last 3 yrs
   * Conditions associated with insulin resistance such as acanthosis nigricans
   * History of vascular disease including heart attack, stroke, angina, coronary heart disease, atherosclerosis, congestive heart failure or peripheral arterial disease

Exclusion Criteria:

* Prior participation in VL-2701
* Receiving investigational treatments in the past 14 days
* Psychosocial issues that interfere with an ability to follow study procedures
* Conditions that cause secondary diabetes including Cushing's syndrome, acromegaly, hemochromatosis, pancreatitis, or cystic fibrosis
* Diagnosed with any type of diabetes, including type 1 or 2
* Taking glucose lowering medications
* Known to be pregnant
* Receiving dialysis or having known renal compromise
* Scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
* Recent (within past month) or current oral steroid therapy or topical steroids applied to the left forearm; inhaled steroid therapy is not excluded Current chemotherapy, or chemotherapy within the past 12 months
* Receiving medications that fluoresce
* Known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)
* Prior bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers age 18 and above, of either sex and of any ethnic background, will be recruited at up to 12 clinical sites. All subjects will be at risk for diabetes based on the American Diabetes Association Standard of Care Guidelines. Those in the 18-44 age group will have an additional risk factor, and the addition of the waist circumference and hypertension thresholds from the National Cholesterol Education Program Adult Treatment Panel III Guidelines for metablolic syndrome
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Validation of SCOUT DS algorithm, ROC performance equivalency to FPG and A1c for detection of abnormal glucose tolerance. | Outcome measure is determined 2-3 months after completion of Visit 3
  The relative true positive and relative true negative fractions between the SCOUT DS and FPG tests for detecting abnormal glucose tolerance (2 hr OGTT value ≥ 140 mg/dL)

SECONDARY OUTCOMES:
Receiver operator characteristic area under the curve, sensitivity, specificity, and postive & negative predictive values of the SCOUT DS, FPG, and A1C tests for detection of abnormal glucose tolerance, and the intra- & inter-day SCOUT DS test | Outcome measure is determined 2-3 months after completion of Visit 3

CONTACTS AND LOCATIONS:
Overall Officials: John Maynard, MS, Study Director — VeraLight, Inc.
Locations (12):
- United States (12):
  - Accelovance - Huntsville, Huntsville, Alabama
  - Accelovance - San Diego, CA, San Diego, California
  - Radiant Research, Inc. - Chicago, Chicago, Illinois
  - Accelovance - Peoria, IL, Peoria, Illinois
  - Radiant Research, Inc. - Kansas City, Kansas City, Kansas
  - Accelovance - Rockville, MD, Rockville, Maryland
  - Radiant Research, Inc. - Minneapolis, Minneapolis, Minnesota
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Radiant Research, Inc. - Cincinnati, Cincinnati, Ohio
  - Juno Research, LLC, Houston, Texas
  - Dynamed Clinical Research, LP, Houston, Texas
  - Radiant Research, Inc. - San Antonio, San Antonio, Texas